CLINICAL TRIAL: NCT06207903
Title: Investigating Participation Behavior: An Observational Study in Mild Cognitive Impairment Clinical Trials
Brief Title: Navigating the Clinical Research Process for Mild Cognitive Impairment
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 58428170
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participation in medical research usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the completion of these specific demographic groups.

This trial will admit a wide range of data on the clinical trial experience of mild cognitive impairment patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future mild cognitive impairment patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of mild cognitive impairment
* Participant must be 18 years of age or older
* Participant must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, and other requirements of the study.

Exclusion Criteria:

* Pregnant or lactating woman
* Participant is actively receiving study therapy in another
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mild cognitive impairment patients who are actively considering participating in a clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a mild cognitive impairment clinical research. | 3 months
Number of mild cognitive impairment study participants who remain in clinical study until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Petersen RC. Mild Cognitive Impairment. Continuum (Minneap Minn). 2016 Apr;22(2 Dementia):404-18. doi: 10.1212/CON.0000000000000313. PMID 27042901
- [Background] Breton A, Casey D, Arnaoutoglou NA. Cognitive tests for the detection of mild cognitive impairment (MCI), the prodromal stage of dementia: Meta-analysis of diagnostic accuracy studies. Int J Geriatr Psychiatry. 2019 Feb;34(2):233-242. doi: 10.1002/gps.5016. Epub 2018 Nov 27. PMID 30370616
- [Background] Chou YH, Sundman M, Ton That V, Green J, Trapani C. Cortical excitability and plasticity in Alzheimer's disease and mild cognitive impairment: A systematic review and meta-analysis of transcranial magnetic stimulation studies. Ageing Res Rev. 2022 Aug;79:101660. doi: 10.1016/j.arr.2022.101660. Epub 2022 Jun 6. PMID 35680080

DOCUMENTS (1):
  • Informed Consent Form (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT06207903/ICF_000.pdf